CLINICAL TRIAL: NCT03992573
Title: The Influence of Concentrated Growth Factors (CGF) Application on Post-operative Complications.
Brief Title: CGF Influence on Post-operative Complications.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: CGF; Bone Loss; Post-operative Wound Healing
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Procedure: CGF application
- Control group (No Intervention)

INTERVENTIONS:
Procedure: CGF application — CGF application into post-operative soft tissue and bone defects
  Arms: Study group

SUMMARY:
The aim of the study is to evaluate the influence of CGF application into post-operative soft tissue and bone defects on post-operative complications and wound healing.

DETAILED DESCRIPTION:
The research was conducted in twenty patients with symmetric single tooth qualified to extraction. On one side of dental arch, post-operative region was field with CGF material, while on the other side it was left to normal healing. In both cases pain, swelling, alveolar osteitis, antibiotics and analgesics intake in post-operative period were evaluated in the first, fourth and seventh day after surgery. Wound healing was assessed seven and thirty days after extraction.

ELIGIBILITY:
Inclusion Criteria:

* no known medical history of abnormal platelet counts,
* patients with symmetric teeth qualified for extraction,

Exclusion Criteria:

* systemic diseases,
* pregnancy,
* lactation,
* drugs known to affect the number or function of platelets,
* abnormal platelet counts

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain vs. CGF application | 24 hours
  In order to evaluate the relationship between intensity of pain after surfery and filling the alveolus with platelet-rich plasma, , NRS (Numeric Rating Scale) pain scale is used.
  NRS scale, ranges from 0 to 10; where 0 refers to no pain and 10 refers to most severe pain.

SECONDARY OUTCOMES:
Occurrence of swelling | 24 hours
  The presence of swelling was evaluated using zero one system.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Surgery, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No